CLINICAL TRIAL: NCT03834649
Title: Evaluation of Soft Tissue Biotype and Volume Stability After Soft Tissue Augmentation by Using Mucograft® Versus Partially De-epithelized Connective Tissue Graft to Enhance the Pontic Site in Single Missing Tooth With Deficient Ridge: Randomized Clinical Trial
Brief Title: Pontic Site Development Using Soft Tissue Augmentation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nouran Abdulla Mater,MD (Other)
Responsible Party: Sponsor-Investigator, Nouran Abdulla Mater,MD, Lectural assistant, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 271188
Record Dates: First submitted 2019-01-22; First posted 2019-02-08 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Mucograft

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mucograft (Active Comparator): Soft tissue augmentation of the defective alveolar ridge using Mucograft inside the prepared vestibular pouch leaving part of the mucograft exposed at the crestal area and will be sutured using 5/0 suture material around the defect margin and secured in the vestibular pouch.
  Interventions: Procedure: Mucograft
- Partially de-epithelialized connective tissue graft (Experimental): Soft tissue augmentation of the defective alveolar ridge using Partially de-epithelialized connective tissue graft by preparing vestibular pouch at the defect site and place the de-epithelialized part inside the pouch leaving the epithelialized part sutured and exposed at the crestal area
  Interventions: Procedure: partially de-epithelized connective tissue graft

INTERVENTIONS:
Procedure: partially de-epithelized connective tissue graft — graft procedures to obtain simultaneous tissue augmentation in the horizontal and vertical dimensions. The donor site was prepared with a full-thickness coronal dissection and a partial-thickness apical dissection.The objectives were to use a single procedure to achieve simultaneously apico-coronal and buccolingual augmentation,to have a smaller open wound in the donor site and less patient discomfort, and to guarantee better revascularization of the onlay section aided by the submerged connective tissue section of the graft.
  Other Names: pontic site development; Combination onlay-inlay grafts
  Arms: Partially de-epithelialized connective tissue graft
Procedure: Mucograft — For preprosthetic defects, a standard mucosal augmentation procedure, which is well reported in the literature, was performed. The surgical site produced by the surgery leaves a "denuded area" supraperiosteally that is addressed by "grafting" with a xenogeneic collagen membrane (Mucograft).
  purpose of the surgery is to improve the quantity of attached mucosa to facilitate the final dental reconstruction
  Other Names: pontic site development; pre-prosthetic development
  Arms: Mucograft

SUMMARY:
in patients with vertical or horizontal defective of there ridge it is difficult to have prosthetic restoration with natural appearance emetating and simulating the adjacent abutment emergence profile so this study aims to develop the defective area using two different materials of soft tissue grafting techniques to restore the missing tissue and regain soft tissue volume and profile

DETAILED DESCRIPTION:
PICO P: single pontic site with deficient ridge. I: Soft tissue augmentation with partially de-epithelized connective tissue graft.

C: Soft tissue augmentation with Mucograft. O: Soft tissue biotype, Soft tissue volume, pain score and patient satisfaction.

Preoperative measures:

* All subjects will pass through phase I therapy (Supragingival scalling, subgingival debridement and oral hygiene instructions) before any surgical procedures.
* After 4 weeks, all subjects will be examined to determine patient compliance with oral hygiene procedures (tooth brushing twice daily and chlorhexidine HCL 1.25% mouthwash twice daily).
* Eligible patients will be randomized before being enrolled in the study. (T-1 +4 weeks)
* Study casts for case study will be fabricated and clinical photographs will be taken.
* Assessment of edentulous defect site and neighboring teeth will be performed by scanning the study casts.

Surgical phase (T0):

The same operator (N M) will perform all procedures under local anesthesia (4% articaine with 1/200 000 adrenaline Solution), using a local infiltration technique.

The recipient site will be prepared using 15c-blad creating a full-thickness coronal dissection and a partial thickness apical dissection creating a vestibular pouch.

The grafting procedure then performed and graft will be fixed by suturing at the periphery of the flap using 5/0 suture material and the rest will be inserted in the vestibular pouch.

The patient will have printed post-surgical instruction and precautions.

* Intervention for control group :

  1. The recipient site will be prepared with a full-thickness coronal dissection and a partial thickness apical dissection to creat a vestibular pouch.
  2. The acellular matrix (Mucograft®) will be sutured using 5/0 suture material around the defect margin and secured in the vestibular pouch.
* Intervention for test group :

  1. The recipient site will be prepared with a full-thickness coronal dissection and a partial thickness apical dissection vestibular pouch.
  2. The graft which is composed of two parts:The coronal part, which is epithelialized

     * The apical part, which is formed of connective tissue only.
  3. On the defect area, the crestal surface is de-epithelialized with a beveled incision and the apical surface is prepared with a partial-thickness dissection with two vertical- releasing incisions extended apically, without involving the adjacent papillae, in order to create a pouch area.
  4. The onlay section (epithelialized area) of the graft will be sutured on the crestal surface of the defect, while the inlay section (connective tissue) will be inserted and secured in the vestibular pouch area.
* Post-operative care:

As with any regenerative site, caution must be exercised in post-operative care and during oral hygiene practices at or near the surgical site. After 12 hours 875 mg of Amoxicillin and 125 mg of Clavulanic acid tablet (1 g Amoxicillin Clavulanate) twice daily for 7 days, anti-inflammatory tablet (Amphiltirne ) if the patient need ,maximum three times/day and chlorhexidine HCL 1.25% mouth wash mouthwash twice daily are prescribed. Sutures will be removed after 14 days. (12)

* Follow-up (T1, T2,T3):

(T1):2 weeks post-operatively sutures removal . (T2) 3 months post-operatively appointments will be assigned for the prosthetic preparation and temporization for 2 weeks (T3): 6 months post-operatively appointments will be assigned for the prosthetic delivery and fill in the Questionnaire.

* Criteria for discontinuing intervention:

  * Infection and sloughing of the graft.
  * if the patient wouldn't commit to the follow-ups.
* Strategies to improve adherence to intervention protocol:

Patient preparation in terms of improving oral hygiene and first phase therapy procedures will be performed for patient to doctor trust. Complete information concerning the protocol will be provided and simplified to the patient with reasoning of all the steps included as the importance of the follow up visits and home medication.

Relevant concomitant care and interventions that are permitted or prohibited during the trial:

Postoperatively the patients will be using analgesics, oral antibiotic therapy, and chlorhexidine HCL 1.25% mouthwash mouthwash for at two week.

ELIGIBILITY:
Inclusion Criteria:

* Single missing tooth and the patient decides to have fixed prosthesis as a treatment option for tooth replacement.
* Horizontal and\or vertical ridge defect at the pontic site
* Sufficient inter-arch distance.
* Restorable neighbouring abutments.
* Periodontally sound abutments.
* Skilled and motivated patient in maintaining good oral hygiene.

Exclusion Criteria:

* Multiple neighboring missing teeth.
* Systemic diseases that could affect treatment outcome.
* Poor oral hygiene.
* Patient is not motivated to have the treatment.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-08-25 (Estimated); Study Completion 2020-09-25 (Estimated)

PRIMARY OUTCOMES:
Soft tissue Biotype (% of the change in soft tissue thickness of keratinized mucosa) | 6 month
  % of the change in soft tissue thickness of keratinized mucosa through Trans mucosal probing by periodontal probe.

SECONDARY OUTCOMES:
soft tissue stability (% of the difference between baseline and post-opertively results through measuring from the crest of edentulous area to Mucogingival line by periodontal prob) | 6 month
  % of the difference between baseline and post-opertively results through measuring from the crest of edentulous area to Mucogingival line by periodontal prob.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt